CLINICAL TRIAL: NCT02897427
Title: Throat and Other HPV-Related Cancers in Men: Identifying Them Early (TRINITY Study)
Brief Title: Throat and Other HPV-Related Cancers in Men: Identifying Them Early
Acronym: TRINITY
Status: Active, not recruiting | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Collaborators: University of Texas Southwestern Medical Center (Other); Cancer Prevention Research Institute of Texas (Other)
Responsible Party: Principal Investigator, Erich Sturgis, Professor and Vice-Chair of Clinical Affairs, Dept of Otolaryngology-Head and Neck Surgery; Brown Foundation Endowed Chair; Head, Neck, & Thyroid Cancer Multidisciplinary Program Director, Baylor College of Medicine
Other Study IDs: BCM H-49215; NCI-2018-02604 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); H-49215 (Other: Baylor College of Medicine)
Record Dates: First submitted 2016-09-07; First posted 2016-09-13 (Estimated); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Human Papillomavirus Infection
Keywords: HPV; HPV-related oropharyngeal cancer; cancer screening; HPV-related cancers
MeSH Terms: conditions — Papillomavirus Infections | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Plasma and Oral Rinse samples will be retained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Screening (specimen collection, HPV testing): STAGE I: Participants fill out a survey and undergo collection of blood and oral rinse samples.
  STAGE II: Participants complete a head and neck exam by using brushing of the oropharyngeal mucosa, a thorough oropharyngeal exam including narrow band imaging, collection of oral rinse sample, transcervical ultrasonography of the neck lymph nodes and oropharynx, anoscopy, penile exam, and complete Papanicolaou/HPV testing. Participants undergo repeat oropharyngeal screening, oral HPV DNA test, oral HPV integration testing, ultrasound, and blood sample collection once every year for 5 years. Select participants will provide oral rinse sample by mail every six months.
  Interventions: Other: Biomarker Analysis; Procedure: Biospecimen Collection; Procedure: Ultrasonography

INTERVENTIONS:
Other: Biomarker Analysis — Complete HPV testing
Procedure: Biospecimen Collection — Undergo collection of blood and oral gargle samples
Procedure: Ultrasonography — Undergo transcervical ultrasonography
  Other Names: 2-Dimensional Grayscale Ultrasound Imaging; 2-Dimensional Ultrasound Imaging; 2D-US; Ultrasound; Ultrasound Imaging; Ultrasound Test; Ultrasound, Medical; US

SUMMARY:
This trial studies the screening of human papillomavirus (HPV)-related oropharyngeal and anogenital cancers. Learning the relationship between HPV and cancer risk in men who test positive for HPV antibodies or circulating HPV DNA may help doctors to develop early methods of screening for certain types of cancer, and screening for HPV may help doctors to learn which patients may be at a higher risk for developing certain types of cancer.

DETAILED DESCRIPTION:
PRIMARY SCIENTIFIC OBJECTIVES:

I. To determine the association of antibodies to human papillomavirus type 16 (HPV16) early (E) antigens and circulating HPV16 DNA (cHPVDNA) with oral HPV16 prevalence.

II. To determine the association of antibodies to HPV16 E antigens and/or cHPVDNA with site-specific HPV16 DNA prevalence, viral persistence, or cellular transformation (cancer and pre-cancer).

III. To determine the association of 12-month persistence of oral rinse HPV16 DNA with site-specific oropharyngeal HPV16 DNA prevalence, viral persistence, or cellular transformation (cancer and pre-cancer).

EXPLORATORY SCIENTIFIC OBJECTIVE:

I. To explore the use of a blood-based point-of-care assay to determine HPV16 E antibody serologic status.

OUTLINE:

STAGE I: Participants undergo collection of blood and oral rinse samples.

STAGE II: Participants complete a head and neck exam with swab of the oropharyngeal mucosa, a thorough oropharyngeal exam including narrow band imaging, collection of oral rinse sample, transcervical ultrasonography of the neck lymph nodes and oropharynx, anoscopy, and complete Papanicolaou/HPV testing. Participants undergo repeat oropharyngeal screening, oral HPV DNA test, oral HPV integration testing, ultrasound, and blood sample collection once every year for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Stage 1 Inclusion Criteria: United States (US) resident
* Stage 1 Inclusion Criteria: Fluent in English
* Stage 1 Inclusion Criteria: Sign an approved informed consent document
* Stage 2 (longitudinal study) Inclusion Criteria:

  * Eligible for and enrolled in Stage 1
  * Test positive to HPV16 E antibodies; be identified as a negative control; test positive for oral HPV16 infection by oral rinse; or test positive for cvDNA
  * Sign an approved informed consent document

Exclusion Criteria:

* Stage 1 Exclusion Criteria: Patients with previously documented squamous cell carcinoma of the oropharynx, anus, or penis
* Stage 1 Exclusion Criteria: Received radiation cancer therapy to the head and neck in the past
* Stage 1 Exclusion Criteria: On active cancer therapy now or in the past 6 months
* Stage 1 Exclusion Criteria: Ever had a transplant (stem cell, bone marrow, or solid organ)
* Stage 1 Exclusion Criteria: Patients who received blood transfusions in the last 6 months
* Stage 1 Exclusion Criteria: Other medical or psychiatric illness or social situation that would limit study compliance
* Stage 2 (longitudinal study) Exclusion Criteria: Any seronegative and cvDNA-negative man who tests negative for oral HPV16 DNA by swab and oral rinse at two consecutive follow-up visits will be excluded from further follow-up. Any man who is seropositive, cvDNA-positive, or has evidence of integration at any time will continue to be followed regardless of oral HPV16 status

Ages: 50 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants willing to have HPV test
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2017-03-28 (Actual); Primary Completion 2027-03-28 (Estimated); Study Completion 2027-03-28 (Estimated)

PRIMARY OUTCOMES:
Cancer detection rate of the seropositive group | Up to 5 years
  Will use the proportion equality test to compare the cancer detection rate of the seropositive group using the screening strategy with the historical rate of 0.08 (4/50). To evaluate the performance of the new techniques for early detection, will test whether the proportion of patients diagnosed at stage I, II, or III from the screening strategy is larger than the historical rate of 17.7% using the proportion equality test. Will further compute and compare the pre-cancer detection rates with the historical information.
Prevalence of serum antibodies to human papillomavirus (HPV)16 E antigens | Up to 5 years
  Will calculate the prevalence of serum antibodies to HPV16 E antigens along with 95% confidence intervals. Will use descriptive statistics to summarize the demographic and sexual behavior characteristics of study participants overall and by HPV16 E antibody status (positive, negative). Logistic regression models will be used to determine the association between serostatus or oral HPV infection status and demographic, socioeconomic, and behavioral factors.

CONTACTS AND LOCATIONS:
Overall Officials: Erich M. Sturgis, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- See also: Baylor College of Medicine Website — https://www.bcm.edu/